CLINICAL TRIAL: NCT03422679
Title: A Phase I/IIA, Multi-Centre, Open-Label, Dose-Escalation Study With Expansion Arms to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CB-103 Administered Orally in Adult Patients With Locally Advanced or Metastatic Solid Tumours and Haematological Malignancies Characterised by Alterations of the NOTCH Signalling Pathway
Brief Title: Study of CB-103 in Adult Patients With Advanced or Metastatic Solid Tumours and Haematological Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: business reason
Sponsor: Cellestia Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB103-C-101
Record Dates: First submitted 2018-01-19; First posted 2018-02-06 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Colorectal Cancer; Adenoid Cystic Carcinoma; Non-hodgkin Lymphoma; Glomus Tumor, Malignant; Hepatocellular Carcinoma; Osteosarcoma; T-ALL
Keywords: advanced solid tumours; haematological malignancies; phase I/II; NOTCH pathway; pan-NOTCH inhibitor
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Carcinoma, Adenoid Cystic; Lymphoma, Non-Hodgkin; Glomus Tumor; Carcinoma, Hepatocellular; Osteosarcoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CB-103 (Experimental): CB-103 capsules will be administered orally in treatment cycles of 28-days each.
  Interventions: Drug: CB-103

INTERVENTIONS:
Drug: CB-103 — Hard gelatine capsules taken orally during treatment period. Treatment cycle is 28 days.

SUMMARY:
This is a phase I/II, non randomized, open-label, dose escalation study to investigate the safety, tolerability and preliminary efficacy of CB-103.

DETAILED DESCRIPTION:
This Phase I/IIA, open label, multicenter, dose escalation study of CB-103 in patients with Locally Advanced or Metastatic Solid Tumours and Haematological Malignancies. After providing signed informed consent, patients will be screened for entry into the study. The study will be conducted in 2 stages: dose escalation in Part A of the study (Phase I) followed by dose expansion in Part B (Phase IIA).

Escalation cohorts will receive repeat doses of CB-103 to determine the MTD and RP2D.

CB-103 will be administered orally in treatment cycles of 28-days each. Aim of the expansion Phase IIA, Part B of the study will be to collect preliminary evidence of anti-tumour activity.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Disease

   * Patients with histologically or cytologically confirmed solid tumours (breast cancer (triple negative breast cancer [TNBC], ER+/-, HER2+/-), gastrointestinal (GI) cancers (resistant to oxaliplatin or irinotecan-based therapy colorectal cancer [CRC]), osteosarcoma, adenoid cystic carcinoma (ACC), and malignant glomus tumour) that are surgically unresectable, locally advanced, or metastatic and whose disease has progressed on at least one line of systemic therapy (with the exception of ACC patients who are allowed to be systemic treatment-naïve) and for whom no established therapeutic alternatives exist. Any other solid cancer (including lymphoma) with a confirmed NOTCH1-4 activating mutation or genetic lesion.
   * Relapsed or refractory (r/r) T-cell acute lymphoblastic leukaemia (T-ALL) or lymphoma (T-LBL) with a confirmed NOTCH pathway activation. Refractory patients are defined as T-ALL/T-LBL patients with ≥ 5% bone marrow blasts, and/or concomitant extramedullary involvement, who have not achieved a CR after standard induction/consolidation therapy attempt.
2. Demography: men and women ≥ 18 years old
3. Adequate organ function and laboratory results
4. Adequate contraceptive measures
5. Signed informed consent

EXCLUSION CRITERIA

1. Medical History

   1. Patients with symptomatic CNS metastases (neurologically unstable or requiring increasing doses of steroids to control their CNS disease)
   2. Hypersensitivity to any of the excipients of CB-103
   3. Patients with unresolved nausea, vomiting, or diarrhoea of CTCAE grade > 1
   4. Impairment of GI function or presence of GI disease that may significantly alter the absorption of CB-103
   5. History of second or other primary cancer with the exception of:

      * Curatively treated non-melanomatous skin cancer
      * Curatively treated cervical cancer or breast carcinoma in situ
      * Other primary solid tumour treated with curative intent and no known active disease present and no treatment administered during the last 2 years.
2. Exclusionary concurrent medical conditions Impaired cardiac function or clinically significant cardiac diseases.
3. Prior Therapy

   * In patients with solid tumours cytotoxic chemotherapy within 3 weeks
   * In T-ALL/T-LBL patients, prior anticancer therapy less than 2 weeks prior to starting therapy or 5 half-lives (whichever is longer) with exceptions.
   * Radiation therapy within 2 weeks of scheduled CB-103 dosing day 1
   * Immunotherapy, biological therapies, targeted small molecules, hormonal therapies within 3 weeks of scheduled CB-103 dosing day 1
   * Unresolved toxicity CTCAE grade > 1 from previous anti-cancer therapy or radiotherapy (excluding neurotoxicity, alopecia, ototoxicity, lymphopenia), or incomplete recovery from previous surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Garalda, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (16):
- United States (3):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson, Houston, Texas
- France (2):
  - Centre Hospitalier Lyon-Sud, Lyon
  - Hôpital Saint-Louis, Paris
- Germany (3):
  - Charite- Universitaetsmedizin Berlin- Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Nationales Centrum für Tumorerkrankungen Heidelberg, Heidelberg
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital - Yonsei Cancer Center, Seoul
- Spain (4):
  - Hospital Quirón Barcelona, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Catalan Institute of Oncology, Barcelona
  - Hospital Ramón y Cajal, Madrid
- Switzerland (2):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Kantonsspital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanna GJ, Stathis A, Lopez-Miranda E, Racca F, Quon D, Leyvraz S, Hess D, Keam B, Rodon J, Ahn MJ, Kim HR, Schneeweiss A, Ribera JM, DeAngelo D, Perez Garcia JM, Cortes J, Schonborn-Kellenberger O, Weber D, Pisa P, Bauer M, Beni L, Bobadilla M, Lehal R, Vigolo M, Vogl FD, Garralda E. A Phase I Study of the Pan-Notch Inhibitor CB-103 for Patients with Advanced Adenoid Cystic Carcinoma and Other Tumors. Cancer Res Commun. 2023 Sep 14;3(9):1853-1861. doi: 10.1158/2767-9764.CRC-23-0333. PMID 37712875
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: CB-103 13mg once daily.
- Cohort 2: CB-103 26mg once daily
- Cohort 3: CB-103 52mg once daily
- Cohort 4: CB-103 104mg once daily
- Cohort 5: CB-103 148mg once daily
- Cohort 6: CB-103 217mg once daily
- Cohort 7: CB-103 348mg once daily
- Cohort 8: CB-103 522mg once daily
- Cohort 9: CB-103 250mg twice daily
- Cohort 10: CB-103 300mg twice daily, 5 days on, 2 days off
- Cohort 11: CB-103 400mg twice daily, 5 days on, 2 days off
- Cohort 12: CB-103 500mg twice daily, 5 days on, 2 days off
- Confirmatory Cohort: CB-103 500mg once daily
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12 | Confirmatory Cohort
Started (Part A - dose escalation was completed. Part B - dose expansion was never opened.) | 5 | 3 | 7 | 7 | 3 | 4 | 3 | 9 | 5 | 6 | 4 | 8 | 15
Completed (Part A - dose escalation was completed. Part B - dose expansion was never opened.) | 5 | 3 | 7 | 7 | 3 | 4 | 3 | 9 | 5 | 6 | 4 | 8 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12 | Confirmatory Cohort | Total
Number analyzed (Participants) | 5 | 3 | 7 | 7 | 3 | 4 | 3 | 9 | 5 | 6 | 4 | 8 | 15 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 5 | 3 | 3 | 2 | 5 | 3 | 5 | 3 | 4 | 12 | 55
  >=65 years | 2 | 0 | 3 | 2 | 0 | 1 | 1 | 4 | 2 | 1 | 1 | 4 | 3 | 24
Age, Continuous [Mean (Full Range); unit: years] | 57.2 [39 to 74] | 55.7 [39 to 74] | 52.7 [25 to 67] | 54.4 [38 to 70] | 51.3 [44 to 62] | 54.8 [41 to 69] | 61.7 [49 to 76] | 56.6 [28 to 76] | 64.6 [56 to 75] | 54 [42 to 72] | 51.5 [23 to 74] | 58.6 [25 to 75] | 46.9 [23 to 71] | 54.4 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 3 | 2 | 2 | 5 | 2 | 4 | 1 | 2 | 5 | 34
  Male | 4 | 2 | 4 | 4 | 0 | 2 | 1 | 4 | 3 | 2 | 3 | 6 | 10 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 5 | 3 | 7 | 7 | 2 | 4 | 3 | 9 | 4 | 6 | 4 | 7 | 9 | 70
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  South Korea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9
  United States | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5 | 3 | 13
  Switzerland | 1 | 2 | 3 | 3 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 15
  Germany | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 5
  Spain | 4 | 1 | 4 | 4 | 3 | 4 | 2 | 5 | 3 | 3 | 0 | 2 | 2 | 37

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Number of patients with dose limiting toxicity during the first cycle.
  DLT is defined as a severe adverse event or abnormal laboratory value assessed as unrelated to disease progression, inter-current illness, or concomitant medications, that occurs ≤ 28 days following the first dose of CB-103 (Cycle 1).
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 12: CB-103 500mg twice daily, 5 days, 2 days off
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12 | Confirmatory Cohort
Number analyzed (Participants) | 5 | 3 | 7 | 7 | 3 | 4 | 3 | 9 | 5 | 6 | 4 | 8 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Overall Response Rate
Description: Number of patients with an overall response rate (CR+PR assessed by RECSIT v1.1 or CR or CRi by NCCN guidelines) up to 24 months
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12 | Confirmatory Cohort
Number analyzed (Participants) | 5 | 3 | 7 | 7 | 3 | 4 | 3 | 9 | 5 | 6 | 4 | 8 | 15
Participants | 1 | 2 | 5 | 5 | 2 | 1 | 2 | 4 | 2 | 5 | 1 | 4 | 3

ADVERSE EVENTS:
Time Frame: From Cycle 1 Day 1 through Safety Follow-up (28 days after the last dose of CB-103), up to 24 months
Description: The occurrence of the adverse events was sought by questioning of the patient at each visit during the study. Adverse events also may be detected when they are volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12 | Confirmatory Cohort
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/7 | 0/7 | 0/3 | 0/4 | 0/3 | 0/9 | 0/5 | 0/6 | 0/4 | 0/8 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/7 | 1/7 | 0/3 | 0/4 | 0/3 | 0/9 | 1/5 | 0/6 | 0/4 | 0/8 | 1/15
Other Adverse Events (participants affected / at risk) | 3/5 | 2/3 | 5/7 | 4/7 | 2/3 | 3/4 | 3/3 | 7/9 | 4/5 | 6/6 | 4/4 | 7/8 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=3) | Cohort 3 (N=7) | Cohort 4 (N=7) | Cohort 5 (N=3) | Cohort 6 (N=4) | Cohort 7 (N=3) | Cohort 8 (N=9) | Cohort 9 (N=5) | Cohort 10 (N=6) | Cohort 11 (N=4) | Cohort 12 (N=8) | Confirmatory Cohort (N=15)
Liver Function Test Increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Steven-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=3) | Cohort 3 (N=7) | Cohort 4 (N=7) | Cohort 5 (N=3) | Cohort 6 (N=4) | Cohort 7 (N=3) | Cohort 8 (N=9) | Cohort 9 (N=5) | Cohort 10 (N=6) | Cohort 11 (N=4) | Cohort 12 (N=8) | Confirmatory Cohort (N=15)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (4)
dyschromatopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 5 (6) | 3 (3) | 3 (4) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 2 (6) | 2 (4) | 2 (8) | 3 (13) | 2 (2)
vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Partners shall provide to Cellestia any proposed publication or oral pesentation relating to the study or the study drug or the results at least 60 days prior to the intended submission or presentation of the publication to allow Cellestia to review it. If Cellestia doesn't provide any comments within the sixty day period, Partner are free to publish.

DOCUMENTS (2):
  • Study Protocol (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03422679/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT03422679/SAP_002.pdf